CLINICAL TRIAL: NCT02907008
Title: Sleep Quality and Risk of Intubation in Intensive Care Units Patients With Hypoxemic Acute Respiratory Failure
Acronym: HIGH SLEEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HIGH SLEEP
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Sleep Quality; Hypoxemic Acute Respiratory Failure; Intubation Risk
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: Polysomnography

SUMMARY:
The aim of the study is to evaluate the impact of sleep quality on intubation rate in intensive care units patients with acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure
* hypoxemia with PaO2/FiO2 ratio < 300 mmHg
* aged of 18 years or more

Exclusion Criteria:

* Need of immediate intubation
* Need of vasopressor drugs
* coma with Glasgow scale < 8
* Acute respiratory failure linked to cardiogenic pulmonary oedema
* Chronic respiratory insufficiency
* Peripheral or central nervous system pathology
* Known psychiatric pathology or agitation
* Patient with decision of no intubation
* Patient refusal
* Pregnant or breastfeeding women
* Patient under legal guardianship or protection
* Patients with no health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care units patients with hypoxemic acute respiratory failure
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
to compare the intubation rate of patients with hypoxemic acute respiratory failure between those who have a poor quality of sleep and those who have a good quality of sleep | 24h

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Poitiers, Poitiers, France